CLINICAL TRIAL: NCT02873546
Title: Evaluation de l'Effet de la tDCS Sur Les Fonctions Cognitives de Patients Souffrant de Maladie d'Alzheimer et Maladies apparentées au Stade léger
Brief Title: tDCS Effect on Cognitive Functions From Patients With Alzheimer's Disease or Progressive Primary Aphasia
Acronym: ALSTICO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Centre Hospitalier Universitaire Dijon (Other); Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: API/2011/24
Record Dates: First submitted 2016-08-11; First posted 2016-08-19 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Alzheimer's Disease; Progressive Primary Aphasia; Early or Mild State
MeSH Terms: conditions — Alzheimer Disease; Pick Disease of the Brain | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- anodal tDCS on left DLPFC (F3) (Active Comparator): tDCS is a non-invasive neuromodulation method, which delivers a constant current of low intensity (1 mA) during 30 minutes for 10 sessions. Anode is placed on the scalp facing on left DLPFC (F3) and cathode between Fp2-F8 EEG-repair.
  Interventions: Device: transcranial Direct Current Stimulation (tDCS)
- sham tDCS on left DLPFC (F3) (Sham Comparator): Sham tDCS differs from active tDCS by the interruption of stimulation after 15 sec and reactivation of the stimulation 15 sec before the end of the session (30 minutes - 10 sessions. Anode is placed on the scalp facing on left DLPFC (F3) and cathode between Fp2-F8 EEG-repair.
  Interventions: Device: transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: transcranial Direct Current Stimulation (tDCS) — After locating the stimulation areas, treatment will be delivered during 30-minute session. Treatment will be occur 2 session per day during 5 consecutive days. Subjects will be monitored during tDCS sessions for any side effects or adverse events.
  Other Names: EldithDC-NeuroConn Stimulator (NeuroConn Gmbh, Germany)

SUMMARY:
The purpose of this study is to evaluate the effect of 10 sessions of anodal transcranial Direct Current Stimulation (tDCS - 1 mA) applied to left Cortex DorsoLateral PreFrontal (CDLPF) of Alzheimer's or Primary Progressive Aphasia (PPA) patients compared to the application of a placebo tDCS (sham procedure) on cognitive functions, which are evaluated at short term (1 week post-treatment) and mild term (3 weeks post-treatment).

After unblinding, patients who received placebo treatment could be received active tDCS.

ELIGIBILITY:
Inclusion Criteria:

* National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINCDS-ADRADA) criteria (Alzheimer's patient) OR Gordo-Tempini criteria (PPA's patient)
* CDR score ≤ 2
* treatment by IAChE ≥ 3 months
* MADRS score < 18
* w/o severe progressive somatic pathology (especially tumor diseases)

Exclusion Criteria:

* last neuropsychological assessment < 6 months
* presence of a specific contraindication for tDCS (e.g. personal history of epilepsy, metallic head implant, cardiac pacemaker)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2013-07-19 (Actual); Primary Completion 2018-01-31 (Estimated); Study Completion 2018-07-31 (Estimated)

PRIMARY OUTCOMES:
change from baseline cognitive functions at 3 weeks | baseline, day 5 and 3 weeks post-tDCS
  neuropsychological assessments include Rapid battery tests (Bereay et al., 2015)

CONTACTS AND LOCATIONS:
Overall Officials: Claire Paquet, MD PhD, Principal Investigator — Assitance Publique - Hôpitaux Paris; Bernard Bonnin, MD PhD, Principal Investigator — Centre Hospitalier Universaitaire Dijon
Locations (3):
- France (3):
  - CHU Besancon - Clinical Psychiatric Department, Besançon
  - Hopital Universitaire Dijon, Dijon
  - Assistance Publique - Hôpitaux Paris, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bereau M, Sylvestre G, Mauny F, Puyraveau M, Baudier F, Magnin E, Berger E, Vandel P, Galmiche J, Chopard G. [Assessment of 10 years of memory consultations in the Franche-Comte: Description and analysis of the RAPID regional database]. Rev Neurol (Paris). 2015 Sep;171(8-9):655-61. doi: 10.1016/j.neurol.2015.04.008. Epub 2015 Jul 23. French. PMID 26212200